CLINICAL TRIAL: NCT05008705
Title: Effects of Protein Intake Plus Neuromuscular Electrical Stimulation on Muscle Mass in Hospitalized Elderly: a Randomized Controlled Clinical Study
Brief Title: Protein Intake Plus Neuromuscular Electrical Stimulation on Muscle Mass in Hospitalized Elderly
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Hamilton Augusto Roschel da Silva, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE43707021.5.0000.0068
Record Dates: First submitted 2021-07-29; First posted 2021-08-17 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Atrophy, Muscular
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients allocated to this arm will be submitted to intervention (protein supplementation plus neuromuscular electrostimulation).
  Interventions: Dietary Supplement: Protein supplementation; Device: Neuromuscular electrostimulation.
- Placebo (Placebo Comparator): Patients allocated to this arm will be submitted to a placebo intervention (isocaloric supplement plus sham for neuromuscular electrostimulation).
  Interventions: Dietary Supplement: Placebo (isocaloric supplement); Device: Sham for neuromuscular electrostimulation.

INTERVENTIONS:
Dietary Supplement: Protein supplementation — Patients will receive diary 2 doses of the protein supplement
  Arms: Intervention
Device: Neuromuscular electrostimulation. — Patients will receive diary sessions of neuromuscular electrostimulation.
  Arms: Intervention
Dietary Supplement: Placebo (isocaloric supplement) — Patients will receive diary 2 doses of the isocaloric supplement
  Arms: Placebo
Device: Sham for neuromuscular electrostimulation. — Patients will not receive neuromuscular electrostimulation.
  Arms: Placebo

SUMMARY:
This study aims to investigate the effects of supplementation of protein plus sessions of electrostimulation on muscle mass, length of hospital stay, readmission and mortality of hospitalized elderly.

DETAILED DESCRIPTION:
Hospitalized elderly people show malnutrition, physical inactivity, and pronounced systemic inflammation which may be exacerbated the catabolic state and promote drastic muscle wasting during the hospitalization and, thus increasing the length of stay, morbidity, and mortality. Therefore, the aim of this study is to investigate the effects of supplementation of protein plus sessions of electrostimulation on muscle mass, length of hospital stay, readmission, and mortality of hospitalized elderly.

ELIGIBILITY:
Inclusion Criteria:

* both sex;
* 65 years and older;
* hospital stay less than 48 hours;

Exclusion Criteria:

* cancer in the last 5 years;
* delirium;
* cognitive deficit that impossibility the patient to read and sign the informed consent form;
* neurological disease;
* neurodegenerative muscular disease;
* impossibility to receive the intervention.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Vastus Lateralis Muscle Cross-sectional Area | From date of admission until the date of medical discharge. Up to 30 days.
  Vastus Lateralis Muscle Cross-sectional Area will be assessed through ultrasound

SECONDARY OUTCOMES:
Muscle function | From date of admission until the date of medical discharge. Up to 30 days.
  Muscle function evaluated trough battery of test
Nutritional status | From date of admission until the date of medical discharge. Up to 30 days.
  Nutritional status will be assessed through nutritional records during hospital stay
Handgrip strength | From date of admission until the date of medical discharge. Up to 30 days.
  Strength will be evaluated using handgrip strength test
Functional independence | From date of admission until the date of medical discharge. Up to 30 days.
  Functional independence will be assessed using Barthel Index
Length of hospital stay | From date of admission until the date of medical discharge. Up to 30 days.
  Length of hospital stay will be the time (in days) until medical discharge.
Mortality | From date of admission until the date of medical discharge. Up to 30 days.
  Mortality rate in percent
Hospital readmission post-medical discharge | 6 months post-medical discharge
  Hospital readmission post-medical discharge will be the number of times that he is admitted in the hospital post-medical discharge.
Health costs | 6 months post-medical discharge
  Health costs will be estimated by means of the questionnaire with questions about the use of health services or equipment.

CONTACTS AND LOCATIONS:
Overall Officials: Hamilton Roschel, PhD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No